CLINICAL TRIAL: NCT02810574
Title: Combining Noninvasive Brain Stimulation and Cognitive Training on Tobacco Craving
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2013-336
Record Dates: First submitted 2016-05-31; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Active noninvasive brain stimulation and cognitive training (Active Comparator): In active condition, subject will receive stimulation during all the 30-minute stimulation period combined with cognitive training.
  Interventions: Behavioral: Cognitive training; Device: Noninvasive brain stimulation (active)
- Sham noninvasive brain stimulation (Sham Comparator): In sham condition, subject will receive stimulation only during the first 30 seconds of the 30-minute stimulation period combined with cognitive training.
  Interventions: Behavioral: Cognitive training; Device: Noninvasive brain stimulation (sham)

INTERVENTIONS:
Behavioral: Cognitive training
Device: Noninvasive brain stimulation (active) — Neuroconn DC-STIMULATOR PLUS
  Arms: Active noninvasive brain stimulation and cognitive training
Device: Noninvasive brain stimulation (sham) — Neuroconn DC-STIMULATOR PLUS
  Arms: Sham noninvasive brain stimulation

SUMMARY:
The purpose of this study is to determine whether combining noninvasive brain stimulation with cognitive training can reduce craving in adults with tobacco use disorder.

ELIGIBILITY:
Inclusion Criteria:

* 20-60 years old
* Smoking > 15 cigarettes per day
* Tobacco Use Disorder according to Diagnostic and Statistical Manual V criteria

Exclusion Criteria:

* Contraindications to noninvasive brain stimulation
* Psychiatric or neurologic condition

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Changes in tobacco craving assessed by the Questionnaire of Smoking Urge | immediately before and immediately after the end of the noninvasive brain stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Interdisciplinaire de Recherche en Réadaptation et Intégration, Québec, Quebec, Canada